CLINICAL TRIAL: NCT04627571
Title: Structural and Functional Changes of Corneal Innervation After Treatment With Cenegermin
Brief Title: Corneal Nerves After Treatment With Cenegermin
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Principal Investigator, Simon Fung, Principal Investigator, University of California, San Francisco
Other Study IDs: 20-000833
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Neurotrophic Keratitis
Keywords: cenegermin; neurotrophic keratopathy; corneal nerve; corneal sensation
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient Population: Patients diagnosed with neurotrophic keratopathy.
  Interventions: Drug: Cenegermin Ophthalmic Solution [Oxervate]

INTERVENTIONS:
Drug: Cenegermin Ophthalmic Solution [Oxervate] — An 8-week course of topical cenegermin eye drops given 6 times daily would be started in the affected eye, in conjunction with the pre-existing medical treatment for neurotrophic keratopathy. Patients will be followed-up at 4 weeks, 6 weeks, 8 weeks, 3 months, 6 months, 9 months and 12 months (±2 weeks at each time point) after treatment. At each visit, patients will be assessed to determine the corneal epithelial defect and corneal sensation.

SUMMARY:
Neurotrophic keratopathy (NK) is a condition in which patients have fewer or complete absence of nerves in the cornea, characterized by the reduced or absent corneal sensation. The lack of nerves in the cornea also result in damages of the cornea and in severe situation the loss of the eye.

Cenegermin (trade name Oxervate) is a nerve growth factor eye drops designed to treat NK, and currently, it is the only FDA-approved medication for this purpose.

Even though cenegermin is effective in the majority of patients, there is a lack of understanding of how cenegermin works in the eye.

In this study, investigators aim to determine the structural and functional effects of cenegermin on the cornea, using non-invasive technologies including in vivo confocal microscopy on study participants with NK over the course of a year.

DETAILED DESCRIPTION:
Cenegermin (OxervateTM) is a recombinant human form of nerve growth factor developed by Dompé Farmaceutici S.p.A. for patients who are diagnosed with corneal epithelial defects due to moderate to severe stages of NK.

ELIGIBILITY:
Inclusion Criteria

1. Patients ≥18 years of age; AND
2. Persistent corneal epitheliopathy that is refractory to treatments for ≥2 weeks; AND
3. Evidence of decreased corneal sensitivity, defined as ≤45mm on Cochet-Bonnet esthesiometer, within the area of the persistent corneal epitheliopathy; AND
4. Evidence of decreased corneal sensitivity, defined as above, in ≥1 corneal quadrant outside the persistent corneal epithelial defect.

Exclusion Criteria

1. Patients with severe neurotrophic keratopathy characterized by corneal stromal ulceration involving over 75% of the total central corneal thickness and impending perforation.
2. Patients who have used cenegermin eyedrops, autologous serum eyedrops, plasma-rich plasma eyedrops, or umbilical cord eyedrops for the treatment of neurotrophic keratopathy 8 weeks prior to study recruitment.
3. Corneal surgery (including keratoplasty or refractive surgical procedures) within three months before study enrollment.
4. Presence of concurrent bacterial or fungal infection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age or older, who have a persistent corneal epitheliopathy due to neurotrophic keratopathy that is refractory to conventional non-surgical treatments for 2 weeks or more, and who fulfill the inclusion and exclusion criteria detailed above.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in corneal nerve fiber density (CNFD) | 1 year
  To determine the changes in corneal nerve fiber density (CNFD), assessed by in vivo confocal microscopy.

SECONDARY OUTCOMES:
Duration of changes in CNFD | 1 year
  To determine the duration of the changes in corneal nerve fiber density (CNFD), assessed by in vivo confocal microscopy.

OTHER OUTCOMES:
Presence/absence of Changes in Dry Eye Symptom | 1 year
  To determine changes in dry eye symptom scores assessed by the Ocular Surface Disease Index in patients initiated on cenegermin for recalcitrant neurotrophic keratopathy. A score ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Changes in Tear Production | 1 year
  To determine the changes in tear production in patients initiated on cenegermin for recalcitrant neurotrophic keratopathy.
Changes in Tear Characteristics | 1 year
  To determine the changes in tear film osmolarity in patients initiated on cenegermin for recalcitrant neurotrophic keratopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacchetti M, Lambiase A. Diagnosis and management of neurotrophic keratitis. Clin Ophthalmol. 2014 Mar 19;8:571-9. doi: 10.2147/OPTH.S45921. eCollection 2014. PMID 24672223
- [Background] Bonini S, Lambiase A, Rama P, Caprioglio G, Aloe L. Topical treatment with nerve growth factor for neurotrophic keratitis. Ophthalmology. 2000 Jul;107(7):1347-51; discussion 1351-2. doi: 10.1016/s0161-6420(00)00163-9. PMID 10889110
- [Background] Lambiase A, Sacchetti M, Bonini S. Nerve growth factor therapy for corneal disease. Curr Opin Ophthalmol. 2012 Jul;23(4):296-302. doi: 10.1097/ICU.0b013e3283543b61. PMID 22543481
- [Background] Bonini S, Lambiase A, Rama P, Filatori I, Allegretti M, Chao W, Mantelli F; REPARO Study Group. Phase I Trial of Recombinant Human Nerve Growth Factor for Neurotrophic Keratitis. Ophthalmology. 2018 Sep;125(9):1468-1471. doi: 10.1016/j.ophtha.2018.03.004. Epub 2018 Apr 10. No abstract available. PMID 29653861
- [Background] Ting DSJ. Re: Bonini et al.: Phase 2 randomized, double-masked, vehicle-controlled trial of recombinant human nerve growth factor for neurotrophic keratitis (Ophthalmology. 2018;125:1332-1343). Ophthalmology. 2019 Feb;126(2):e14-e15. doi: 10.1016/j.ophtha.2018.09.017. No abstract available. PMID 30683186
- [Background] Pflugfelder SC, Massaro-Giordano M, Perez VL, Hamrah P, Deng SX, Espandar L, Foster CS, Affeldt J, Seedor JA, Afshari NA, Chao W, Allegretti M, Mantelli F, Dana R. Topical Recombinant Human Nerve Growth Factor (Cenegermin) for Neurotrophic Keratopathy: A Multicenter Randomized Vehicle-Controlled Pivotal Trial. Ophthalmology. 2020 Jan;127(1):14-26. doi: 10.1016/j.ophtha.2019.08.020. Epub 2019 Aug 26. PMID 31585826
- [Background] Mastropasqua L, Lanzini M, Dua HS, D' Uffizi A, Di Nicola M, Calienno R, Bondi J, Said DG, Nubile M. In Vivo Evaluation of Corneal Nerves and Epithelial Healing After Treatment With Recombinant Nerve Growth Factor for Neurotrophic Keratopathy. Am J Ophthalmol. 2020 Sep;217:278-286. doi: 10.1016/j.ajo.2020.04.036. Epub 2020 May 6. PMID 32387431
- See also: Related Info — https://link.springer.com/article/10.1007/s40135-020-00228-y